CLINICAL TRIAL: NCT01155622
Title: Pilot Randomized Clinical Trial Comparing the Efficacy of Two Different Hypothermia Temperatures for Treatment of Comatose Patients Recovered From an Out-of-hospital Cardiac Arrest
Brief Title: Trial of Different Hypothermia Temperatures in Patients Recovered From Out-of-hospital Cardiac Arrest
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Esteban Lopez de Sa Areses, MD, FESC, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hypothermia_32vs34
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Non-environmental Hypothermia; Cardiac Arrest
Keywords: Hypothermia, induced; Cardiac arrest; Disability evaluation; Cardiac arrhythmia; Ventricular function; Internal cooling; Out-of-hospital cardiac arrest; Post-cardiac arrest syndrome
MeSH Terms: conditions — Heart Arrest; Hypothermia; Arrhythmias, Cardiac; Out-of-Hospital Cardiac Arrest; Post-Cardiac Arrest Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 32º Celsius (Active Comparator): Endovascular Cooling was set at a target temperature of 32°C
  Interventions: Procedure: Endovascular Cooling
- 34º Celsius (Active Comparator): Endovascular Cooling was set at a target temperature of 32°C
  Interventions: Procedure: Endovascular Cooling

INTERVENTIONS:
Procedure: Endovascular Cooling — Infusion of <8°C cold saline followed by the implantation of the Icy 9.3F 38-cm catheter (ZOLL Medical Corporation, Chelmsford, MA) placed in the inferior vena cava through a femoral vein connected to the Thermogard XP Temperature Management System (ZOLL Medical Corporation). Cooling was set at a maximum rate with a target temperature of 32°C or 34°C according to randomization.

SUMMARY:
Mild therapeutic hypothermia in the temperature range of 32º - 34ºC. improves survival in patients recovered from a ventricular fibrillation cardiac arrest. The same therapy is suggested with less evidence for asystole as first rhythm after cardiac arrest. The purpose of this study is to determine whether different temperature targets (32º vs 34º) may have different efficacy in the treatment of post-cardiac arrest patients. If successful, this pilot study will eventually form the basis for a larger, multicentric randomized clinical trial.

DETAILED DESCRIPTION:
Patients admitted consecutively were potentially eligible for the study if they had a witnessed out-off hospital cardiac arrest (OHCA) apparently related to heart disease and an interval of <60 minutes from collapse to return of spontaneous circulation (ROSC). Additional inclusion criteria were:

1. Age >18 years.
2. Initial registered rhythm of a shockable rhythm (ventricular fibrillation or pulseless ventricular tachycardia) or asystole.

Exclusion criteria were:

1. Known pregnancy
2. Glasgow Coma Scale score after ROSC >8.
3. Cardiogenic shock (a systolic blood pressure of <80 mm Hg despite inotrope infusion >30 minutes).
4. Other nonshockable rhythms (pulseless electric activity).
5. Terminal illness present before the OHCA.
6. Possible causes of coma other than cardiac arrest (drug overdose, head trauma, or cerebrovascular accident).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Resuscitated patients from a cardiac arrest with first rhythm of ventricular fibrillation or asystole
* Witnessed cardiac arrest
* Estimated delay between cardiac arrest and advanced resuscitation < 20 min.
* Resuscitation time from first contact to recovery of spontaneous circulation < 60 min.
* Hemodynamic stability (Mean blood pressure [BP] >60 mmHg), with or without inotropic drugs, before randomization
* Glasgow coma score <9 without sedation before randomization

Exclusion Criteria:

* Pregnant women or suspected pregnancy or fertile women without a negative pregnancy test
* Suspected non-cardiac arrest caused coma
* Electrical instability (uncontrollable life-threatening arrhythmias)
* Hemodynamic instability (Mean BP ≤60 mmHg), refractory to volume infusion or inotropic drugs
* Refractory hypoxemia (saturation <85% with FiO2=100%)
* Previous known terminal illness
* Active bleeding or known coagulopathy
* Opposition from patient's family to enter the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-03; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Survival free from severe dependence (Barthel index <60) | 6 months

SECONDARY OUTCOMES:
Survival at 6 months | 6 months
Barthel Index at 6 months | 6 months
Life threatening arrhythmias in different hypothermia temperatures | 48 hours (during hypothermia)
  New life-threatening arrhythmias during hypothermia: ventricular fibrillation, sustained (>30 sec.) monomorphic or polymorphic ventricular tachycardia, extreme bradycardia (heart rate <35 bpm. and/or pauses >3 sec.)
Impact on ventricular function of different hypothermia temperatures | 48 hours During hypothermia
  Echocardiographic evaluation of possible impact of different hypothermia temperatures on ventricular diastolic and systolic function

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Lopez-de-Sa, MD, FESC, Principal Investigator — Intensive Cardiac Care Unit. Department of Cardiology. Hospital Universitario La Paz
Locations (1):
- Intensive Cardiac Care Unit. Hospital Universitario la Paz, Madrid, Madrid, Spain

REFERENCES:
- [Result] Lopez-de-Sa E, Rey JR, Armada E, Salinas P, Viana-Tejedor A, Espinosa-Garcia S, Martinez-Moreno M, Corral E, Lopez-Sendon J. Hypothermia in comatose survivors from out-of-hospital cardiac arrest: pilot trial comparing 2 levels of target temperature. Circulation. 2012 Dec 11;126(24):2826-33. doi: 10.1161/CIRCULATIONAHA.112.136408. Epub 2012 Nov 6. PMID 23136160